CLINICAL TRIAL: NCT04831619
Title: Contribution of PET Scans for the Preoperative Assessment of Symptomatic Endometriosis Lesions: TEP-ENDORUN
Brief Title: Contribution of PET (Positron Emission Tomography) Scans for the Preoperative Assessment of Symptomatic Endometriosis Lesions: TEP-ENDORUN
Acronym: TEP-ENDORUN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/CHU/12
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET scanner in addition to MRI (Experimental)
  Interventions: Drug: PET scanner with injection of 18 FDG (18F-2-fluoro-2-deoxy-D-glucose) (radiolabel)

INTERVENTIONS:
Drug: PET scanner with injection of 18 FDG (18F-2-fluoro-2-deoxy-D-glucose) (radiolabel) — A PET scan will be performed in the patients included, in addition to the conventional imaging workup (MRI, endovaginal and pelvic ultrasound).

SUMMARY:
Endometriosis is an inflammatory condition that is often treated by surgery. MRI and ultrasound are used for the preoperative morphological assessment. Currently, only surgery allows the exhaustive and qualitative diagnosis of lesions.

The PET scan, fixing in certain inflammatory pathologies and in certain cases of endometriosis, could refine this assessment by evaluating the location of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 and under 50
* Patient with symptomatic endometriosis with indication for surgery
* Showing at least one typical endometriosis lesion on MRI, greater than 5mm
* Accepting surgical management
* Having signed an informed consent after information
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient who has received an injection with GnRH (gonadotropin-releasing hormone ) analogues for less than 3 months (because it induces the quiescence of the disease which is no longer stimulated by estrogen secretion)
* Patient with a history of heavy abdominopelvic surgery
* Diabetic patient
* Patient unable to understand the interest of the study
* Patient already included in another therapeutic trial with an experimental molecule.
* Persons referred to in articles L1121-5 to L1121-8 of the PHC (public health code) (corresponding to all protected persons: pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, minor, and person making the subject to a legal protection measure: guardianship or curators)
* Contraindications to PET Scanner (major claustrophobia, contraindication or hypersensitivity to 18-FDG or one of its excipients, contraindication or hypersensitivity to Ultravist® or one of its excipients, etc.)
* Contraindication to surgery or anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the PET scan in the diagnosis of endometriosis lesions compared to surgery in terms of number of lesions diagnosed and locations. | at inclusion (before surgery)
  Total number of endometriosis lesions diagnosed by the PET scanner

SECONDARY OUTCOMES:
Compare the results of the PET scanner and MRI for the sensitivity of detection of endometriosis lesions | up to 14 weeks (after surgery)
  number of endometriosis lesions
Compare the results of the PET scanner and MRI for the sensitivity of detection of endometriosis lesions | up to 14 weeks (after surgery)
  location of endometriosis lesions
Define a reading threshold of SUV (Standardized Uptake Value) on a PET scanner for the diagnosis of endometriosis | up to 14 weeks (after PET-Scanner)
  degree of inflammation of the cells

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire Réunion, Saint-Denis
  - CHU de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No